CLINICAL TRIAL: NCT04479826
Title: Unannounced Meal Handling of Advanced Closed Loop Insulin Delivery in Monitored Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Prof. Amir Tirosh, Clinical Professor, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sheba-19-5955-at-ctil
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: Advanced hybrid closed loop system — Free living follow-up of meal handelling

SUMMARY:
The study will follow participants for the periods of 3 months while using an advanced hybrid closed loop algorithm in free living conditions . Each period will have a different meal handling protocols. The objective is to identify the mitigation of the algorithm with different meal handling approaches.

ELIGIBILITY:
1. Subject is 20 to 70 years of age at time of screening
2. Subject's weight is between 50 and 120 kg
3. A clinical diagnosis of Type 1 diabetes as determined by the Investigator for a minimum of 36 months prior to enrollment
4. Subject has ongoing use of an insulin pump and rtCGM ≥ 6 months prior to screening
5. Subject has an A1C value ≤ 10.0% demonstrated at the time of enrollment.
6. Subject uses a rapid-acting analogue insulin in his/her pump
7. Patient is willing to undergo all study procedures
8. English proficiency
9. Minimum daily insulin requirement (Total Daily Dose) of greater than or equal to 8 units

Exclusion:

1. Female subject who has a positive serum pregnancy screening test, or who plans to become pregnant during the course of the study
2. Subject has unresolved adverse skin condition, or unable to tolerate tape adhesive, in the area of sensor placement or device replacement (e.g., psoriasis, rash, Staphylococcus infection)
3. Subject has a history of hypoglycemic seizure or hypoglycemic coma within the past 12 months
4. Subjects currently taking adjunct therapy with SGLT2-inhibitors, GLP-1 mimetics, Amylin.
5. Subject has a history of seizure disorder unrelated to diabetes within the past 12 months
6. Gastroparesis, uncontrolled thyroid disorder, Addison dis. , Pituitary insufficiency
7. Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), congestive heart failure, ventricular rhythm disturbances, or thromboembolic disease within the past 6 months
8. Subject has a presence of a cardiac pacemaker or any other device that may be sensitive to radio frequency telemetry
9. Subject has any condition, including screening lab values that in the opinion of the Investigator may preclude him/her from participating in the study and completing study related procedures
10. Subject is actively participating in other investigational study (drug or device)
11. Subjects who consume alcohol daily

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Time in ranges | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shalit R, Minsky N, Laron-Hirsh M, Cohen O, Kurtz N, Roy A, Grosman B, Benedetti A, Tirosh A. Unannounced Meal Challenges Using an Advanced Hybrid Closed-Loop System. Diabetes Technol Ther. 2023 Sep;25(9):579-588. doi: 10.1089/dia.2023.0139. PMID 37335759